CLINICAL TRIAL: NCT06600282
Title: A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Parecoxib After Intravenous Bolus of Parecoxib in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence of Two Formulations of Parecoxib in Healthy Volunteers Under Fasting Conditions
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: YSP-RQH3001-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Pain; Bioequivalence Study in Healthy Subjects
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, balanced, two-treatment, two-period, two-sequence, single dose, two-way crossover study under fasting conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reference Drug (Active Comparator): Active Ingredient: Parecoxib Dosage Form: Lyophilized powder for injection Strength: 40 mg/vial Dose: 40 mg (single intravenous bolus)
  Interventions: Drug: Parecoxib
- Test Drug (Experimental): Active Ingredient: Parecoxib Dosage Form: Lyophilized powder for injection Strength: 40 mg/vial Dose: 40 mg (single intravenous bolus)
  Interventions: Drug: Parecoxib

INTERVENTIONS:
Drug: Parecoxib — Pharmacokinetic study under fasting conditions

SUMMARY:
A randomized, single-dose, two-way crossover study to evaluate bioequivalence of two formulations of parecoxib after intravenous bolus of parecoxib in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects between 20-45 years of age (inclusive) at the screening visit.
2. Body mass index (BMI) between 18 and 27 kg/m2 (not inclusive) at the screening visit.
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in Electrocardiogram (ECG) results within six months prior to Period I dosing.
   * no particular clinical significance in general disease history within two months prior to Period I dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes Alanine aminoTransferase (ALT), Aspartate aminoTransferase (AST), gamma-GT, alkaline phosphatase, total bilirubin, albumin, glucose, Blood urea nitrogen (BUN), uric acid, creatinine, total cholesterol, and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials, and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes pH, blood, glucose, ketones, bilirubin, and protein.
7. Subjects must use an acceptable method of birth control (e.g. abstinence, condom, intrauterine device, and vasectomy) for the duration of the study.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, urinary tract, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease.
2. A clinically significant illness or surgery within four weeks prior to Period I dosing.
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime.
6. History of alcohol addiction or abuse within last five years.
7. History of allergic response(s) to parecoxib, valdecoxib or any other related drugs.
8. Evidence of chronic or acute infectious diseases.
9. Positive result for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Female subjects demonstrating a positive pregnancy screen.
11. Female subjects who are currently breastfeeding.
12. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to Period I dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone, and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone, and ranitidine.
13. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu and COVID-19 vaccination) within two weeks prior to Period I dosing.
14. Use of any investigational drug (excluding COVID-19 vaccination) within four weeks prior to Period I dosing.
15. Use of any COVID-19 vaccine within seven days prior to Period I dosing.
16. Donating more than 250 mL of blood within two months prior to Period I dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to Period I dosing.
17. Any other medical reason as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0 (pre-dose), 2, 5, 10, 20, 30, 40, 50 mins, and 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, 24, and 36 hours post dose (a total of 19 samples per subject in one period)
Area under the concentration-time curve from time zero to time of last quantifiable | 0 (pre-dose), 2, 5, 10, 20, 30, 40, 50 mins, and 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, 24, and 36 hours post dose (a total of 19 samples per subject in one period)
Area under the concentration-time curve from time zero to infinity (AUC 0-∞) | 0 (pre-dose), 2, 5, 10, 20, 30, 40, 50 mins, and 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12, 24, and 36 hours post dose (a total of 19 samples per subject in one period)

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan